CLINICAL TRIAL: NCT00696787
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Pregabalin-Referenced, Parallel-Group, Adaptive Design Study of DVS SR in Adult Female Outpatients With Fibromyalgia Syndrome
Brief Title: A Study Evaluating Desvenlafaxine Sustained Release (DVS SR) in Adult Female Outpatients With Fibromyalgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A4-2003
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): In the first stage, subjects were randomly assigned to receive placebo. Study was stopped after stage 1 by sponsor.
  Interventions: Drug: Placebo
- DVS SR (Experimental): In the first stage, subjects were randomly assigned to receive DVS SR 200 mg/day. Study was stopped after stage 1 by sponsor.
  Interventions: Drug: Desvenlafaxine Sustained Release (DVS SR)
- Pregabalin (Active Comparator): In the first stage, subjects were randomly assigned to receive Pregabalin 450 mg/day. Study was stopped after stage 1 by sponsor.
  Interventions: Drug: Lyrica® (Pregabalin)

INTERVENTIONS:
Drug: Desvenlafaxine Sustained Release (DVS SR)
  Arms: DVS SR
Drug: Lyrica® (Pregabalin)
  Arms: Pregabalin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if DVS SR is safe and effective in the treatment of pain associated with fibromyalgia syndrome, and if so to identify the efficacious doses.

ELIGIBILITY:
Inclusion Criteria:

- Fibromyalgia diagnosed according to 1990 American College of Rheumatology criteria

Exclusion Criteria:

* Unstable medical or psychological conditions that would compromise the subject's safety or put the subject at greater risk during study participation
* Other painful conditions that may confound the diagnosis or assessment of fibromyalgia
* Treatment with other drugs for fibromyalgia with 14 days of study start or during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (25):
- United States (25):
  - Huntsville, Alabama
  - Roseville, California
  - San Diego, California
  - Santa Ana, California
  - Walnut Creek, California
  - Jacksonville, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Rockville, Maryland
  - Lansing, Michigan
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Middleton, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the United States from June 2006 to November 2008.
Pre-assignment Details: After a 7 to 30 day screening period, eligible subjects entered a 7 day single blind placebo run-in period during which placebo responses were assessed.
Period: Overall Study
Arm/Group | Placebo | DVS SR | Pregabalin
Started | 40 | 42 | 43
Completed | 25 | 22 | 17
Not Completed | 15 | 20 | 26
Not completed — Adverse Event | 1 | 0 | 6
Not completed — Discontinuation by Sponsor | 9 | 13 | 14
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Failed to return | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DVS SR | Pregabalin | Total
Number analyzed (Participants) | 40 | 42 | 43 | 125
Age Continuous [Mean (Standard Deviation); unit: years] | 46.90 (12.65) | 47.83 (10.53) | 45.42 (12.11) | 46.70 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 43 | 125
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Numeric Rating Scale (NRS)
Description: The primary efficacy variable was the change from baseline on the NRS. The primary time point was the average pain score during the last data-analysis-interval of week 8. The baseline score was the average of the NRS scores across the last 7 days of the screening period (just prior to the start of the placebo run-in). The primary efficacy variable was the pain severity score measured on an 11 point NRS on which 0=no pain and 10=worst possible pain.
Time Frame: Baseline and 8 weeks
Population: The Modified Intent to Treat (MITT) population included all randomized subjects who had taken at least one dose of double-blind test article, who had a baseline primary efficacy evaluation, and who had at least one primary efficacy evaluation on double-blind therapy.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | DVS SR | Pregabalin
Number analyzed (Participants) | 40 | 42 | 43
units on scale | -1.98 (0.37) | -1.60 (0.37) | -1.70 (0.38)
Statistical Analysis 1: Comparison: Placebo vs DVS SR; Test type: Superiority or Other; p = 0.471, ANCOVA; Adjusted mean = -0.38, 95% CI 2-sided [-1.42 to 0.66]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p = 0.604, ANCOVA; Adjusted mean = -0.28, 95% CI 2-sided [-1.33 to 0.77]

2. Secondary Outcome: Change From Baseline on the Numeric Rating Scale (NRS) in the Treatment of Pain Associated With Fibromyalgia in Adult Female Outpatients
Description: The efficacy variable was the change from baseline on the numeric rating scale (NRS). The time point was the average pain score during the last data-analysis-interval of week 8, data analysis interval. The baseline score was the average of the NRS scores across the last 7 days of the screening period (just prior to the start of the placebo run-in). The efficacy variable was the pain severity score measured on an 11 point NRS on which 0=no pain and 10=worst possible pain.
Time Frame: Baseline and 8 weeks
Population: All randomized subjects who had taken at least one dose of double-blind test article, had a baseline primary efficacy evaluation, and had at least one primary efficacy evaluation on double-blind therapy. Subjects who did not complete the study due to its discontinuation were excluded.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Placebo | DVS SR | Pregabalin
Number analyzed (Participants) | 31 | 29 | 29
units on scale | -2.00 (0.37) | -1.64 (0.39) | -1.45 (0.40)
Statistical Analysis 1: Comparison: Placebo vs DVS SR; Test type: Superiority or Other; p = 0.510, ANCOVA; Adjusted mean = -0.35, 95% CI 2-sided [-1.42 to 0.71]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p = 0.317, ANCOVA; Adjusted mean = -0.55, 95% CI 2-sided [-1.64 to 0.54]

ADVERSE EVENTS:
Arm/Group | Placebo | DVS SR | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42 | 1/43
Other Adverse Events (participants affected / at risk) | 25/40 | 25/42 | 32/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | DVS SR (N=42) | Pregabalin (N=43)
Pregnancy and spontaneous abortion (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | DVS SR (N=42) | Pregabalin (N=43)
Eye disorders general (Eye disorders) | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 4 | 6 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 5
Injury, poisoning and procedural complications general (Injury, poisoning and procedural complications) | 2 | 1 | 3
Metabolism and nutrition disorders general (Metabolism and nutrition disorders) | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 16
Headache (Nervous system disorders) | 4 | 2 | 5
Migraine (Nervous system disorders) | 2 | 0 | 1
Somnolence (Nervous system disorders) | 4 | 2 | 6
Insomnia (Psychiatric disorders) | 4 | 1 | 0
Reproductive system and breast disorders general (Reproductive system and breast disorders) | 2 | 0 | 0
Respiratory, thoracic and mediastinal disorders general (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Skin and subcutaneous tissue disorders general (Skin and subcutaneous tissue disorders) | 0 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.